CLINICAL TRIAL: NCT00080847
Title: Standard Dose Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) and Rituximab, or Rituximab and G3139 Phosphorothioate Oligonucleotide (BCL-2 Antisense - NSC-683428) Therapy for Young Patients (< Age 60) With Advanced Stage Diffuse Large B-Cell NHL of Low and Low-Intermediate IPI Risk
Brief Title: S0349 Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone With or Without Oblimersen in Treating Patients With Advanced Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03031; S0349; U10CA032102 (NIH); CDR0000356049 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — oblimersen; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

ARMS (2):
- Arm I (closed to accrual as of 9/21/04) (Experimental): Patients receive rituximab IV over 6 hours, cyclophosphamide IV over 15-45 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1 and oral prednisone on days 1-5.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive oblimersen IV continuously on days 1-7; rituximab IV over 6 hours, cyclophosphamide IV over 15-45 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 5; and oral prednisone on days 5-10.
  Interventions: Biological: oblimersen sodium; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
  Arms: Arm II
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying rituximab and combination chemotherapy to see how well they work compared to oblimersen, rituximab, and combination chemotherapy in treating patients with advanced diffuse large B-cell non-Hodgkin's lymphoma. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of anticancer drugs by making cancer cells more sensitive to the drugs. Combining rituximab and combination chemotherapy with oblimersen may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 1-year progression-free survival probability rate in younger patients with low and low-intermediate IPI risk advanced stage diffuse large B-cell NHL treated with 8-cycles of CHOP-rituximab. (The CHOP-rituximab arm of this study was permanently closed, effective 10/15/04.) II. To estimate the 1-year progression-free survival probability rate in younger patients with low and low-intermediate IPI risk advanced stage diffuse large B-cell NHL treated with 8 cycles of CHOP-rituximab-G3139.

III. To evaluate response (complete, complete unconfirmed, and partial) and toxicity for these regimens in this patient population. (The CHOP-rituximab arm of this study was permanently closed, effective 10/15/04.) IV. To estimate the 1-year progression-free survival and response rate in the subset of patients overexpressing bcl-2 protein.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age-adjusted International Prognostic Index (0 vs 1). Patients are randomized to 1 of 2 treatment arms. (Arm I closed to accrual as of 9/21/04.)

ARM I (closed to accrual as of 9/21/04): Patients receive rituximab IV over 6 hours, cyclophosphamide IV over 15-45 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1 and oral prednisone on days 1-5.

ARM II: Patients receive oblimersen IV continuously on days 1-7; rituximab IV over 6 hours, cyclophosphamide IV over 15-45 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 5; and oral prednisone on days 5-10.

In both arms, treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have previously untreated stage III, IV, or bulky stage II diffuse large B-cell non-Hodgkin's lymphoma which is positive for CD20
* Adequate sections from the original diagnostic specimen must be available for submission for review; an adequate biopsy requires sufficient tissue to establish the architecture and a REAL or WHO histologic subtype with certainty; thus, core biopsies, especially multiple core biopsies MAY be adequate; whereas, needle aspirations or cytologies are not adequate

  * Patients may also be registered to SWOG-8947 and SWOG-8819
* Patients must have an age-adjusted International Prognostic Index score of 0 or 1
* All patients must have bidimensionally measurable disease documented within 28 days prior to registration; patients with non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within 42 days prior to registration
* Patients must have a unilateral bone marrow aspirate and biopsy performed within 42 days prior to registration
* Patients must have a CT scan of the chest and abdomen/pelvis performed within 28 days prior to registration
* Patients must not have clinical evidence of central nervous system involvement by lymphoma; any laboratory or radiographic tests performed to assess CNS involvement must be negative within 42 days of registration
* Patients must not have a previous diagnosis of indolent lymphoma (histologic transformation are ineligible); as patients with nodal diffuse large ell lymphoma may have bone marrow involvement with small lymphocytes, such patients are eligible
* Patients must not have received prior chemotherapy, radiation, or antibody therapy for lymphoma
* All patients must have a Zubrod performance status of 0-2
* Serum LDH must be measured within 28 days prior to registration
* Patients must have a cardiac ejection fraction >= 45% by MUGA scan or an ECHO with no significant abnormalities within 42 days prior to registration
* Patients known to be HIV positive, or who have a history of solid organ transplantation are ineligible as the biology and natural history of HIV associated, or post transplant lymphomas are very different than that of de novo diffuse large cell lymphomas; patients at high risk of hepatitis B virus infection should be screened before initiation of rituximab
* Patients requiring continuing supplemental oxygen therapy are ineligible
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Pregnant or nursing women may not participate due to the potential for congenital abnormalities, and of harm to nursing infants due to this treatment regimen; women or men of reproductive potential may no participate unless they have agreed to use an effective contraceptive method
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday 4 weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
1 year PFS | At 1 year

SECONDARY OUTCOMES:
Overall survival | Up to 7 years
Response | Up to 7 years
1-year PFS in patients who are bcl2+ | At 1 year
Overall survival in patients who are bcl2+ | Up to 7 years
Response in patients who are bcl2+ | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bernstein, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States